CLINICAL TRIAL: NCT06441396
Title: Comparison of the Effects of Telerehabilitation and Video Fundamentals of Exercise on Physical Performance and Body Composition in Older Adult Individuals
Brief Title: Comparison of Telerehabilitation and Video Basics and Exercise in Older Adult Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Özgün Elmas, Research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Hacettepe University-Ftr-Oe
Record Dates: First submitted 2024-05-18; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Tele-rehabilitation; Exercise; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Telerehabilitation is a group Video-based rehabilitation is the other group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Active Comparator): It is a group that performs the given exercise program mutually with the physiotherapist via video connection.
  Interventions: Other: Telerehabilitation
- Video-based rehabilitation (Active Comparator): This is the group that does the given exercises by watching the video.
  Interventions: Other: Video-based rehabilitation (VTR)

INTERVENTIONS:
Other: Telerehabilitation — In the study, the VTR guru was given video footage of 15 exercises previously recorded on camera. The individuals in this group were made to do the exercises together online via the WhatsApp program. Exercises in both groups were planned for 6 weeks, 3 days a week, 25-45 minutes. The main program consists of 15 calisthenic exercises involving the lower extremity, upper extremity and trunk large muscle groups. Exercises in both groups were planned for 6 weeks, 3 days a week, 25-45 minutes. The number of repetitions of each exercise started with 10 and was increased by 5 repetitions every two weeks until it reached 20 repetitions.
  Arms: Telerehabilitation
Other: Video-based rehabilitation (VTR) — In the study, the VTR guru was given video footage of 15 exercises previously recorded on camera. Participants were asked to exercise by watching these videos. In addition, these individuals were interviewed once a week to check the progress of the exercise program. Video images were sent to the intervention group for informational purposes, and the individuals in this group were made to do the exercises together online via the WhatsApp program.
  Arms: Video-based rehabilitation

SUMMARY:
Researchers could not find a study in the literature examining the effectiveness of different technological methods in exercise practices in older adults. Based on this, the aim of this study is to compare the effect of exercise intervention using telerehabilitation and video-based rehabilitation method on physical performance, muscle mass, fat percentage and body mass index.

DETAILED DESCRIPTION:
Telerehabilitation is defined as the use of information and telecommunication technologies to provide healthcare services over a long distance between a patient and a healthcare professional. It involves a multi-component approach such as remote monitoring, e-learning and tele-coaching. The American Telemedicine Association defines telerehabilitation as "the delivery of rehabilitation services through information and communication technologies." It also states that telerehabilitation encompasses a range of rehabilitation and habilitation services, including assessment, monitoring, prevention, intervention, supervision, education, counseling and counseling.

In cases where access to healthcare services is limited, it is recommended to use telerehabilitation to provide effective rehabilitation services to patients. Telerehabilitation is an emerging field that is growing rapidly and becoming an important part of telemedicine and e-health. It is hypothesized that it may offer new possibilities to deliver intervention strategies across the continuum of rehabilitation and that the distance barrier can be minimized to increase access. Minimizing the distance barrier can be achieved through various modes of telecommunications, including voice, video and virtual reality.

Telerehabilitation refers to services provided by occupational therapists, speech therapists, and physical therapists. It provides continuity of service throughout the entire rehabilitation cycle, including assessment, intervention, consultation and education, and has emerged as an effective support for providing home rehabilitation care to recently discharged patients. In the practice of telerehabilitation, it is assumed that patients have various advantages in many respects, as they have the opportunity to perform rehabilitation in their own social environment, can avoid transportation problems, can personally arrange their exercise hours, and are encouraged to self-manage their disease.

The use of telerehabilitation can promote standardization, improve patient compliance with exercise programs, and reduce costs. Additionally, this type of technology can also facilitate participation in rehabilitation when patients cannot access traditional physical therapy services due to geographic challenges or inability to travel.

A Cochrane review found that the technologies used in telerehabilitation interventions were well accepted by patients, but further studies were needed to increase the evidence base for clinical benefits.

Participation in exercise is low in elderly individuals, and the Covid 19 pandemic has further reduced the low participation of the elderly in exercise. For this reason, telerehabilitation for the elderly is becoming more and more important day by day.

Researchers could not find a study in the literature examining the effectiveness of different technological methods in exercise practices in older adults. Based on this, the aim of this study is to compare the effect of exercise intervention using telerehabilitation and video-based rehabilitation method on physical performance, muscle mass, fat percentage and body mass index.

Location of the research: Hacettepe University Faculty of Physical Therapy and Rehabilitation Geriatric Rehabilitation Unit and Lokman Hekim University

Population of the study, sample, research group: The minimum number of participates required to be included in the study was determined by power analysis. It is planned to include individuals applying to Hacettepe University Faculty of Physical Therapy and Rehabilitation Geriatric Rehabilitation Unit and Lokman Hekim University to participate in the research. Individuals who give their written consent and meet the inclusion criteria will be included in the study.

Study design:

Signed consent was obtained from the participants who agreed to participate in the research, and the research was conducted by the researchers within the framework of the ethical rules determined according to the Declaration of Helsinki.

The researchers followed the instructions in the CONSORT checklist used in randomized controlled trials while writing the article.

Individuals over 65 years old who participated in the study were divided into 2 groups (TR and VTR) by computer-generated randomization (allocation ratio of 1:1). The researchers sent only videotaped exercises to the VTR group and were asked to follow the exercises in the videos.

In order to better understand the exercises, the researchers sent these recorded videos to the TR group, and the researchers also had the participants do the exercises online with the help of TR using the WhatsApp program. Before and after the intervention, the participants were evaluated by the researchers in terms of physical performance, muscle mass, fat ratio and BMI. These evaluation results were compared within and between groups. The exercises performed by both participant groups were performed for 25-45 minutes, 3 days a week for 6 weeks.

Both participates groups were given the same exercises.

ELIGIBILITY:
Inclusion Criteria:

* Not having cognitive problems
* Being over 65 years old
* Volunteering to participate in the study

Exclusion Criteria:

* Amputees
* Those who cannot communicate adequately
* Having a neurological or orthopedic problem that will affect functionality
* Those who cannot walk independently
* Those who underwent surgery
* Those with endoprosthesis

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-01-31 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Physical performance tests- 30 seconds chair stand test: | six weeks
  It is performed to evaluate lower extremity endurance. The individual is asked to fully stand up from a chair without armrests and sit back down for 30 seconds. The exact number of standing up and sitting down during thirty seconds is recorded. An increase in the number of starts means better endurance
Physical performance tests- 30 seconds chair stand test-Time up & go test (TUG): | six weeks
  Time up & go test (TUG): It is used to evaluate balance and functional mobility. The person is seated on a chair without armrests, then the person is asked to get up from the chair, walk 3 m, return to the chair and sit down. The time it takes to complete the test is recorded. Decreasing test completion time means better performance
Physical performance tests- Single leg stance: | six weeks
  Single leg stance: Without shoes, they stand on one leg with their hands on their hips, one knee bent, and time is kept. It is performed 3 times for each extremity, the best score is recorded (16).
Physical performance tests- Six-minute walk test: | six weeks
  It is used to determine the functional exercise capacities of participants. Participants are asked to walk quickly for 6 minutes. The distance walked during this time is measured in meters. Long distance indicates better physical performance

SECONDARY OUTCOMES:
Assessing the participants' height | six weeks
  Researchers measure the participants' height using a meter. This recorded value in meters (m) will then be entered into the Inboby 120 device, which gives the participant's weight in kilograms (kg) to the researchers with the help of electrodes.
Evaluation of body mass index | six weeks
  Inbody 120 device shows the participant's body mass index Muscle mass (kg), fat percentage (%) and Body Mass Index (BMI) (kg/m²) values of the participants were measured with the InBody 120 (Biospace, California, USA) bioimpedance analyzer. The device analyzes via tetra polar bio-electrical impedance (BIA). The measurement frequency is between 20-100 kHz. Electric currents pass more easily through body tissues where there is a lot of water (such as blood, urine and muscles) than through other tissues (such as bone, fat or air). With this method, the speed and strength of electrical currents passing through the body are measured and these results are used to determine information such as height, weight, gender and body composition of the person.
Evaluation of height | six weeks
  Inbody 120 device shows the participant's general body weight. Muscle mass (kg), fat percentage (%) and Body Mass Index (BMI) (kg/m²) values of the participants were measured with the InBody 120 (Biospace, California, USA) bioimpedance analyzer. The device analyzes via tetra polar bio-electrical impedance (BIA). The measurement frequency is between 20-100 kHz. Electric currents pass more easily through body tissues where there is a lot of water (such as blood, urine and muscles) than through other tissues (such as bone, fat or air). With this method, the speed and strength of electrical currents passing through the body are measured and these results are used to determine information such as height, weight, gender and body composition of the person.
Evaluation of muscle mass | six weeks
  Inbody 120 device shows the participant's muscle mass. Muscle mass (kg), fat percentage (%) and Body Mass Index (BMI) (kg/m²) values of the participants were measured with the InBody 120 (Biospace, California, USA) bioimpedance analyzer. The device analyzes via tetra polar bio-electrical impedance (BIA). The measurement frequency is between 20-100 kHz. Electric currents pass more easily through body tissues where there is a lot of water (such as blood, urine and muscles) than through other tissues (such as bone, fat or air). With this method, the speed and strength of electrical currents passing through the body are measured and these results are used to determine information such as height, weight, gender and body composition of the person.
Evaluation of fat ratio | six weeks
  Inbody 120 device shows the participant's ratio. Muscle mass (kg), fat percentage (%) and Body Mass Index (BMI) (kg/m²) values of the participants were measured with the InBody 120 (Biospace, California, USA) bioimpedance analyzer. The device analyzes via tetra polar bio-electrical impedance (BIA). The measurement frequency is between 20-100 kHz. Electric currents pass more easily through body tissues where there is a lot of water (such as blood, urine and muscles) than through other tissues (such as bone, fat or air). With this method, the speed and strength of electrical currents passing through the body are measured and these results are used to determine information such as height, weight, gender and body composition of the person.

OTHER OUTCOMES:
Evaluation of muscle strength | six weeks
  Muscle strength was evaluated with a digital dynamometer for the deltoideus-anterior and quadricepsfemoris muscles. The tests were repeated three times on the right and left sides for each muscle, and the average of the three evaluations was recorded in Newtons (N). Jamar hand dynamometer recommended by the American Hand Therapists Association was used to evaluate hand grip strength. Hand grip strength was measured in a sitting position, with the shoulder in adduction and neutral rotation, the elbow in 90 degrees of flexion, the forearm in the middle position and supported, and the wrist in neutral. During the test, 3 measurements were made for hand grip, with a one-minute break between each measurement, and the average was recorded).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elmas O, Cemali M, Livanelioglu A. Comparison of the effects of video conference and video-based home exercise on physical performance and body composition in older adult individuals. Medicine (Baltimore). 2024 Nov 1;103(44):e40329. doi: 10.1097/MD.0000000000040329. PMID 39495999